CLINICAL TRIAL: NCT07277335
Title: Association Between Neuromuscular Variables and Competitive Performance in Weightlifting: an Observational Study With Mexican Athletes [The Kraft Project]
Brief Title: Neuromuscular Variables and Performance in Mexican Weightlifters
Acronym: KRAFT
Status: Recruiting | Type: Observational
Sponsor: Ángel Rodríguez (Network)
Responsible Party: Sponsor-Investigator, Ángel Rodríguez, Researcher, Dynamical Business and Science Society - DBSS International SAS
Organization: Dynamical Business and Science Society - DBSS International SAS (Network)
Other Study IDs: Kraft2025_DBSS; Kraft2025_DBSS (Other: Innovation MX DBSS)
Record Dates: First submitted 2025-11-26; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Isometric Muscle Strength; Jumping Performance; Weightlifting; Performance Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior weightlifters younger than 15 years old
  Interventions: Other: Isometric start position pull (ISPP); Other: Vertical impulse; Other: Performance
- Elite weightlifters older than 18 years old (up to 23 years)
  Interventions: Other: Isometric start position pull (ISPP); Other: Vertical impulse; Other: Performance

INTERVENTIONS:
Other: Isometric start position pull (ISPP) — The participants' force production capacity will be assessed. The test will be conducted on a force platform. Each athlete will perform general and specific warm-up and familiarization with three isometric attempts with CJ grip (~50%, 80% and 100% perceived effort). For measurement, each participant will execute two 3-s maximum attempts with CJ grip, with 1 minute rest between efforts.
Other: Vertical impulse — A force platform will be used to measure the lower-limbs vertical impulse during a The Deep Squat Jump (DSJ). Participants will execute the DSJ without any countermovement, ensuring maintenance of the full squat position for 3-4 seconds before takeoff to avoid any contribution from elastic energy storage.
Other: Performance — Performance indicators will be obtained from official competition records, extracting the best valid loads in Snatch (SN), Clean & Jerk (CJ), and Total (TOT)

SUMMARY:
This study aims to determine whether, within each weight and sex category, higher isometric pull force or greater vertical jump impulse is associated with better final placement in the competition.

DETAILED DESCRIPTION:
This cross-sectional observational study will be conducted during the 2025 "El Pavo" National Tournament, held in San Luis Potosí, Mexico, with athletes officially registered with the Mexican Weightlifting Federation (FMLP). Vertical jump impulse will be assessed using the Deep Squat Jump (DSJ) approximately two hours after each athlete's last valid attempt, followed by the Isometric Pull Start Position (IPSP) test to measure isometric pull force. Competitive performance data-best Snatch (SN), Clean & Jerk (CJ), and Total (TOT)-will be obtained from official competition records, along with the athlete's final placement within their sex and body mass category.

The study will analyze athletes from two age groups (U-15 and Over-18) and both sexes, selecting one light and one heavy body mass division per group. The included divisions are: U-15, Female: -44 kg (light), -63 kg (heavy) and Male: -56 kg (light), -79 kg (heavy); Over-20, Female: -53 kg (light), -77 kg (heavy) and Male: -65 kg (light), -94 kg (heavy)

ELIGIBILITY:
Inclusion Criteria:

* Weightlifters younger than 15 years old and older than 18 years old (up to 23 years), registered to compete in the 2025 "El Pavo" National Tournament with no declared health issues.

Exclusion Criteria:

* Weightlifters registered for the 2025 "El Pavo" National Tournament who present any declared health issues.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Weightlifters younger than 15 years old and older than 18 years old (up to 23 years), who will participate in the 2025 edition of the annual national tournament "El Pavo," organized by the Mexican Weightlifting Federation, will be evaluated
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Isometric start position pull (ISPP) | <5 minutes
  The participants' force production capacity will be assessed. The test will be conducted on a force platform
Vertical impulse | <5 minutes
  A force platform will be used to measure the lower-limbs vertical impulse during a The Deep Squat Jump (DSJ)
Performance | <1 minutes
  The final placement of each athlete in their category

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Bonilla, Study Director — Research Division, Dynamical Business & Science Society-DBSS International SAS; Rodrigo D Merlo, PhD, Study Chair — Research Division, Dynamical Business & Science Society-DBSS International SAS; Ángel Rodríguez-Chávez, Mg, Principal Investigator — Research Division, Dynamical Business & Science Society-DBSS International SAS; Jorge L Petro, Study Chair — Research Division, Dynamical Business & Science Society-DBSS International SAS; Leoncio Moreno, Study Chair — Federación Mexicana de Levantamiento de Pesas; Shyam Chavda, Study Chair — London Sports Institute, Middlesex University, West Stand, Stone X Stadium, Greenlands Lane, London NW4 1RL, UK; Marcos A Soriano, Study Chair — Centre for Sport Studies, Rey Juan Carlos University, 28943 Madrid, Spain; miguel.delolmo@urjc.es
Locations (1):
- Hotel María Dolores, San Luis Potosí City, San Luis Potosí, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joffe SA, Chavda S, Gilham J, Sandercock GRH, Tallent J. A comparison of maximal isometric force in the first pull, transition and second pull of the clean and their contribution to predict performance in national and international level weightlifters. Sports Biomech. 2025 Jan 30:1-17. doi: 10.1080/14763141.2025.2458478. Online ahead of print. PMID 39882780
- [Background] Soriano MA, Flores FJ, Alonso-Aubin DA, Garcia-Sanchez C, Ceniza-Villacastin JA, Jimenez-Ormeno E, Lama-Arenales J, Comfort P. Associations Between Maximum Isometric Strength and Weightlifting Performance in Youth Weightlifters. J Strength Cond Res. 2025 May 1;39(5):570-578. doi: 10.1519/JSC.0000000000005052. PMID 40266638
- [Background] Vizcaya FJ, Viana O, del Olmo MF, Acero RM. Could the deep squat jump predict weightlifting performance? J Strength Cond Res. 2009 May;23(3):729-34. doi: 10.1519/JSC.0b013e3181a04dc3. PMID 19387408